CLINICAL TRIAL: NCT02019745
Title: Effects of Tobacco Products on Live Attenuated Influenza Virus (LAIV) Infections in Human Volunteers
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); Tobacco Centers of Regulatory Science (TCORS (Unknown)
Responsible Party: Sponsor
Other Study IDs: 13-2246; P50HL120100-01 (NIH)
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Influenza, Human; Smoking; Respiratory Tract Infections; Habits
Keywords: Live attenuated influenza virus (LAIV); Flu vaccine; FluMist; Smokers; New and emerging tobacco products
MeSH Terms: conditions — Influenza, Human; Smoking; Respiratory Tract Infections; Habits | interventions — FluMist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine, nasal lavage fluid, nasal epithelial cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LAIV (FluMist): All subjects will receive a 0.2 mL dose of LAIV (FluMist) once during the study.
  Interventions: Biological: LAIV

INTERVENTIONS:
Biological: LAIV — Standard dose of LAIV administered by a licensed health care providers.
  Other Names: FluMist

SUMMARY:
Chronic exposure to (cigarette smoke) CS causes biological changes, including airway remodeling and changes in baseline gene expression profiles at the level of the epithelium. Our own data indicate that chronic exposure to CS suppresses the ability of epithelial cells to enhance antiviral gene expression in response to influenza infection and activate host defense responses. While there is a large body of evidence supporting the notion that exposure to CS causes significant changes in host defense responses, which may be linked to permanent changes in epithelial cells at the genomic level, it is not known whether new and emerging tobacco products have similar or distinct effects.

Using live attenuated influenza virus (LAIV) inoculation in human volunteers, this study will compare influenza-induced responses in non-smokers (NS), cigarette smokers (CS), e-cigarette smokers (EC), hookah smokers (HS), and Little Cigar smokers (LCS) in vivo. This will be done by analyzing nasal viral titers, antiviral defense responses, inflammatory mediator production, and markers of immune responses for LAIV-induced responses between the different groups of volunteers.

DETAILED DESCRIPTION:
Cigarette smoke (CS), e-cigarette smoke (EC), hookah smoke (HS), and Little Cigar smoke (LCS)-exposed populations will be stratified based on their responses to a smoking diary, protocol questionnaire, as well as urine cotinine levels (which should be present in all three groups). We are aware that many current smokers are poly-tobacco product users (i.e. smoke cigarettes in addition to non-cigarette products), which could be confounding our observations. This will be controlled for by having potential volunteers complete a smoking diary and provide daily urine samples for 1 week prior to enrolling in the study. Based on this diary, subjects will be grouped as CS (cigarettes only), EC (e-cigarette smokers and smoking less than ½ pack of cigarettes per week), HS (hookah smokers and smoking less than ½ pack of cigarettes per week), and LCS (little cigar smokers and smoking less than ½ pack of cigarettes per week). Individuals with mixed exposures that exceed those described above (i.e. smoking more than ½ pack of cigarettes per week in addition to smoking hookah, e-cigarettes, or Little Cigars) will be excluded from the studies. Potential subjects will then complete a questionnaire regarding their smoking history, and will undergo urine collection for measurement of cotinine for 7 consecutive days. Subjects will be assigned to the different groups as followed: Group NS (no routine exposure to tobacco smoke, and average log10 urine cotinine/creatinine ratio < 1.0), Group CS (active cigarette smoker and log10 urine cotinine/creatinine ratio > 4), Group EC (active e-cigarette smokers and average log10 urine cotinine/creatinine ratio 1-4), Group HS (active routine hookah smokers and average log10 urine cotinine/creatinine ratio 1-4), or Group LCS (active routine Little Cigars smoker and average log10 urine cotinine/creatinine ratio 1-4).

Study protocol outline:

Screening visit (2-4 weeks prior to Day 0): Obtain informed consent, history (including smoke exposure questionnaire), physical examination, vital signs (VS), blood draw (for anti-influenza antibody titer, HIV and T cell stimulation with flu antigen), urine (for cotinine), nasal lavage (NL, for differential cell count, viral culture and antigen detection, cytokine panel), nasal epithelial lining fluid (ELF, collected with filter paper for cytokine analysis), nasal epithelial biopsy (NB) #1, pregnancy test for females of child bearing potential. In addition, smokers will undergo spirometry.

Subjects will return to the research lab daily the for the week prior to D0 to provide a urine sample for cotinine. Subjects will given a daily smoking/exposure diary during this time to continue throughout the study.

Day 0 (Monday): Obtain VS, NL, ELF, urine. Administer FluMist.

Day 1 (Tuesday): Obtain VS, NL, ELF, urine, NB #2

Day 2 (Wednesday): Obtain VS, NL, ELF, urine

Day 8 +/- 1 day (Monday-Wednesday): Obtain VS, NL, ELF, urine, NB #3

Day 21 +/- 7 days: Obtain VS, blood draw, collect completed smoking/exposure diary

ELIGIBILITY:
Inclusion Criteria:

* Healthy, young nonsmoking adults age 18-45 years who are not routinely exposed to environmental tobacco smoke
* Healthy, young adults age 18-45 years who are active regular smokers (will be stratified based on cigarette, hookah, and Little Cigars)

Exclusion Criteria:

* Pregnancy or nursing;
* history of egg allergy;
* history of allergic rhinitis;
* aspirin therapy;
* asthma;
* immunodeficiency (HIV or other);
* on immunosuppressive drugs including corticosteroids;
* history of Guillain-Barre Syndrome;
* smokers with a forced expiratory volume in 1 second (FEV1) less than 75% predicted at screen;
* Chronic obstructive pulmonary disorder (COPD), cardiac disease, or any chronic cardiorespiratory condition;
* febrile and/or respiratory illness within past 3 weeks prior to entry into study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Nonsmokers
  2. Cigarette smokers
  3. Primarily e-cigarette smokers
  4. Primarily hookah smokers
  5. Primarily Little Cigar smokers
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in nasal responses of nonsmokers (NS), cigarette smokers (CS), e-cigarette smokers (EC), hookah smokers (HS), and Little Cigar smokers (LCS) to live attenuated influenza virus | Baseline, 7 weeks
  Influenza hemagglutinin (HA) messenger ribonucleic acid (mRNA) (normalized to β-actin) will be measured in nasal lavage fluid (NLF) cells from NS, CS, EC, HS, and LCS by quantitative real time-polymerase chain reaction (qRT-PCR) after LAIV inoculation.

SECONDARY OUTCOMES:
Compare smoking (CS, EC, HS, and LCS) and nonsmoking groups (NS) for changes in numbers and activation of inflammatory and immune cells in NLF at specific time points compared to baseline | Basline, 7 weeks
Compare smoking (CS, EC, HS, and LCS) and nonsmoking groups (NS) for change in cytokines/chemokines and other mediators in NLF compared to baseline | Baseline, 7 weeks
  Cytokines and chemokines and other mediators to be measured include, but are not limited to, interferon gamma-induced protein (IP)-10, interleukin (IL)-6, IL-1beta, interferon (IFN)-alpha, IFN-beta, IFN-gamma, tumor necrosis factor (TNF)alpha, IL-8, RANTES, eotaxins, prostaglandin E2 (PGE2), eosinophil cationic protein (ECP), and myeloperoxidase (MPO).
Compare smoking (CS, EC, HS, and LCS) and nonsmoking groups (NS) for changes in influenza-specific antibody production in NLF and serum | Baseline, 7 weeks
  Immunoglobulin (Ig)A will be analyzed in NLF while IgG and IgM will be analyzed in the serum.
Compare smoking (CS, EC, HS, and LCS) and nonsmoking groups (NS) for changes in mucus composition | Basline, 7 weeks
Compare smoking (CS, EC, HS, and LCS) and nonsmoking groups (NS) for genomic signatures induced in epithelial cells | Baseline, 7 weeks
Compare smoking (CS, EC, HS, and LCS) and nonsmoking groups (NS) for epigenomic signatures induced in epithelial cells | Baseline, 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Jaspers, PhD, Principal Investigator — University of North Carolina-Chapel Hill, Dept of Pediatrics
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Rebuli ME, Glista-Baker E, Hoffman JR, Duffney PF, Robinette C, Speen AM, Pawlak EA, Dhingra R, Noah TL, Jaspers I. Electronic-Cigarette Use Alters Nasal Mucosal Immune Response to Live-attenuated Influenza Virus. A Clinical Trial. Am J Respir Cell Mol Biol. 2021 Jan;64(1):126-137. doi: 10.1165/rcmb.2020-0164OC. PMID 33095645